CLINICAL TRIAL: NCT06153238
Title: A Randomized, Double-blind, Parallel-group Study to Compare Pharmacokinetics of GME751 (Proposed Pembrolizumab Biosimilar) and US-licensed and EU Authorized Keytruda® in Participants With Stage II and III Melanoma Requiring Adjuvant Treatment With Pembrolizumab
Brief Title: A PK Study to Compare GME751 (Proposed Pembrolizumab Biosimilar) and US-licensed and EU-authorized Keytruda® in Participants With Stage II and III Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGME751A12101
Record Dates: First submitted 2023-10-11; First posted 2023-12-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GME751 (Experimental): Subjects will receive GME751 via intravenous (IV) infusion.
  Interventions: Drug: GME751
- Keytruda - EU (Active Comparator): Subjects will receive Keytruda-EU via intravenous (IV) infusion.
  Interventions: Drug: Keytruda - EU
- Keytruda - US (Active Comparator): Subjects will receive Keytruda-US via intravenous (IV) infusion.
  Interventions: Drug: Keytruda - US

INTERVENTIONS:
Drug: GME751 — 400 mg Q6W, i.v. infusion, over 24 weeks period
  Arms: GME751
Drug: Keytruda - EU — 400 mg Q6W, i.v. infusion, over 24 weeks period
  Arms: Keytruda - EU
Drug: Keytruda - US — 400 mg Q6W, i.v. infusion, over 24 weeks period
  Arms: Keytruda - US

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic (PK) similarity and efficacy, safety, and immunogenicity of GME751 compared with Keytruda® (pembrolizumab) in subjects with resected advanced melanoma requiring adjuvant treatment with pembrolizumab.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 1:1:1 ratio to receive either GME751, Food and Drug Administration (FDA)-licensed pembrolizumab (Keytruda-US) or European Union (EU)-authorized pembrolizumab (Keytruda-EU). The maximum study duration for a participant will be approximately 28 weeks including screening.

Treatment duration is 24 weeks (4 treatment cycles, each of 6 weeks duration). However, subject should discontinue study participation in case of disease recurrence, unacceptable toxicity or other reasons.

Participants who are benefiting from treatment with pembrolizumab without signs of recurrence or unacceptable toxicity will be eligible for continued pembrolizumab treatment via most suitable option based on the respective country regulations.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Advanced Melanoma
* Completely removed melanoma by surgery performed within 13 weeks of randomization
* Adequate organ function
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Known history or evidence of ocular or uveal melanoma
* Known history of hypersensitivity (grade ≥3) to pembrolizumab or its excipients
* Known History of auto-immune disease
* Received live vaccine ≤30 days before the first study treatment
* Prior treatment with anti-PD-1 agents or agent against another stimulatory or co-inhibitory T cell receptor
* Active autoimmune disease that has necessitated chronic systemic treatment within 2 years before the first study treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve from Time Zero to 42 Days (AUC0-42d) | Day 1 (Postdose) through Day 42
  The PK similarity (AUC0-42d) of GME751 compared with pembrolizumab will be demonstrated in subjects with advanced melanoma in the adjuvant setting.
Area Under the Serum Concentration-time Curve Over the Dosing Interval at Steady State | Week 19 through Week 24
  The PK similarity (AUCtau_ss) of GME751 compared with pembrolizumab will be demonstrated in subjects with advanced melanoma in the adjuvant setting.

CONTACTS AND LOCATIONS:
Locations (61):
- United States (3):
  - Sandoz Investigational Site, Orange, California
  - Sandoz Investigational Site, Clermont, Florida
  - Sandoz Investigational Site, Orange City, Florida
- Bosnia and Herzegovina (4):
  - Sandoz Investigational Site, Banja Luka
  - Sandoz Investigational Site, Mostar
  - Sandoz Investigational Site, Sarajevo
  - Sandoz Investigational Site, Tuzla
- Brazil (12):
  - Sandoz Investigational Site, Barretos
  - Sandoz Investigational Site, Belo Horizonte
  - Sandoz Investigational Site, Canoas
  - Sandoz Investigational Site, Caxias do Sul
  - Sandoz Investigational Site, Curitiba
  - Sandoz Investigational Site, Florianópolis
  - Sandoz Investigational Site, Fortaleza
  - Sandoz Investigational Site, Itajaí
  - Sandoz Investigational Site, Porto Alegre
  - Sandoz Investigational Site, Porto Velho
  - Sandoz Investigational Site, Salvador
  - Sandoz Investigational Site, São José do Rio Preto
- France (2):
  - Sandoz Investigational Site, Besançon
  - Sandoz Investigational Site, Nantes
- Georgia (2):
  - Sandoz Investigational Site, Batumi
  - Sandoz Investigational Site, Tbilisi
- Germany (3):
  - Sandoz Investigational Site, Mainz
  - Sandoz Investigational Site, Münster
  - Sandoz Investigational Site, Tübingen
- Italy (2):
  - Sandoz Investigational Site, Catanzaro
  - Sandoz Investigational Site, Rozzano
- Lithuania (2):
  - Sandoz Investigational Site, Klaipėda
  - Sandoz Investigational Site, Vilnius
- Malaysia (6):
  - Sandoz Investigational Site, George Town
  - Sandoz Investigational Site, Johor Bahru
  - Sandoz Investigational Site, Kuala Lumpur
  - Sandoz Investigational Site, Kuching
  - Sandoz Investigational Site, Malacca
  - Sandoz Investigational Site, Putrajaya
- Mexico (4):
  - Sandoz Investigational Site, Mexico City
  - Sandoz Investigational Site, Oaxaca City
  - Sandoz Investigational Site, San Luis Potosí City
  - Sandoz Investigational Site, Veracruz
- Sandoz Investigational Site, Chisinau, Moldova
- Sandoz Investigational Site, Skopje, North Macedonia
- Sandoz Investigational Site, Bacolod, Philippines
- Romania (2):
  - Sandoz Investigational Site, Bucharest
  - Sandoz Investigational Site, Cluj-Napoca
- Serbia (3):
  - Sandoz Investigational Site, Belgrade
  - Sandoz Investigational Site, Kamenitz
  - Sandoz Investigational Site, Niš
- South Africa (2):
  - Sandoz Investigational Site, Johannesburg
  - Sandoz Investigational Site, Phoenix
- Spain (9):
  - Sandoz Investigational Site, Badalona
  - Sandoz Investigational Site, Barcelona
  - Sandoz Investigational Site, Cáceres
  - Sandoz Investigational Site, Madrid
  - Sandoz Investigational Site, Murcia
  - Sandoz Investigational Site, Santiago de Compostela
  - Sandoz Investigational Site, Seville
  - Sandoz Investigational Site, Valencia
  - Sandoz Investigational Site, Zaragoza
- Turkey (Türkiye) (2):
  - Sandoz Investigational Site, Ankara
  - Sandoz Investigational Site, Yüreğir

IPD SHARING:
Plan to Share IPD: No